CLINICAL TRIAL: NCT00777959
Title: A Phase II Randomized, Placebo Controlled Clinical Trial to Study the Efficacy and Safety of Bicalutamide With or Without Deforolimus (Ridaforolimus) in Men With Asymptomatic, Metastatic Castrate-resistant Prostate Cancer
Brief Title: Bicalutamide and Ridaforolimus in Men With Prostate Cancer (MK-8669-002)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Collaborators: Ariad Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 8669-002; 2008_572
Record Dates: First submitted 2008-10-21; First posted 2008-10-22 (Estimated); Last update posted 2015-08-19 (Estimated); Status verified 2015-08

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — ridaforolimus

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Open Label (Experimental): ridaforolimus (MK8669)+ bicalutamide
  Interventions: Drug: open-label ridaforolimus (MK8669)
- Ridaforolimus (Experimental): ridaforolimus (MK8669)+ bicalutamide
  Interventions: Drug: ridaforolimus (MK8669)
- Placebo (Placebo Comparator): Placebo + bicalutamide
  Interventions: Drug: Comparator: Placebo

INTERVENTIONS:
Drug: ridaforolimus (MK8669) — Three 10 mg tablets administered daily for 5 consecutive days each week followed by 2 days without ridaforolimus and one 50 mg tablet of bicalutamide administered once daily for 7 days each week. Treatment will continue until disease progression.
  Other Names: AP23573
  Arms: Ridaforolimus
Drug: Comparator: Placebo — Three tablets of matching placebo to ridaforolimus administered daily for 5 consecutive days each week followed by 2 days without matching placebo and on 50 mg tablet of bicalutamide administered once daily for 7 days each week. Treatment will continue until disease progression.
  Arms: Placebo
Drug: open-label ridaforolimus (MK8669) — Single dose of three 10 mg tablets ridaforolimus on Day 1, and 50 mg bicalutamide once daily starting on Day 2. On Day 8, patients will begin taking three 10 mg tablets of ridaforolimus daily for 5 consecutive days each week followed by 2 days without ridaforolimus and one 50 mg tablet of bicalutamide once daily for 7 days each week. Treatment will continue until disease progression.
  Other Names: AP23573
  Arms: Open Label

SUMMARY:
This study will look to see if the combination of ridaforolimus and bicalutamide works better than placebo and bicalutamide in men with prostate cancer.

DETAILED DESCRIPTION:
Ridaforolimus (MK8669/AP23573) was also known as deforolimus until May 2009.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed adenocarcinomas of the prostate.
* Evidence of metastatic disease
* Evidence of disease progression including one of the following: increasing levels of PSA, progressive lymph node disease, or worsening bone scan
* PSA level is greater or equal to 7 ng/ml.
* ECOG performance status less than or equal to 1

Exclusion Criteria :

* Previously received bicalutamide, flutamide, or nilutamide within the past 12 months (except for a period of use less than 30 days long).
* Prior chemotherapy for prostate cancer
* Prior rapamycin or rapamycin analogs, including ridaforolimus, everolimus, or temsirolimus.
* Patient is receiving an opioid or narcotic analgesic for pain due to prostate cancer
* Patient has pain related to prostate cancer that warrants the initiation of chemotherapy

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2008-10; Primary Completion 2011-05 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
30% Prostate specific antigen (PSA) decline within 12 weeks | 12 weeks
Number of dose limiting toxicities (DLTs) | Day 1 to Day 35

SECONDARY OUTCOMES:
Prostate specific antigen (PSA) response rate | 12 weeks
Number of patients with progression free survival (PFS) | 12 weeks
Time to prostate specific antigen (PSA) progression | 12 weeks
Pharmacokinetics Maximum Concentration (Cmax), Time to Maximum Plasma Concentration (Tmax), Area Under the Concentration Versus Time Curve (AUC) of Ridaforolimus | 30 Minutes to 24 hour postdose

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Result] Meulenbeld HJ, de Bono JS, Tagawa ST, Whang YE, Li X, Heath KH, Zandvliet AS, Ebbinghaus SW, Hudes GR, de Wit R. Tolerability, safety and pharmacokinetics of ridaforolimus in combination with bicalutamide in patients with asymptomatic, metastatic castration-resistant prostate cancer (CRPC). Cancer Chemother Pharmacol. 2013 Oct;72(4):909-16. doi: 10.1007/s00280-013-2250-6. Epub 2013 Aug 7. PMID 23921574